CLINICAL TRIAL: NCT07344077
Title: Comparison of Radiographic and Functional Outcomes of Minimal Invasive Distal Metatarsal Osteotomy Using 1 Versus 2 Kirshner Wire Fixation in Patients With Severe Hallux Valgus: A Randomized Controlled Trial
Brief Title: Comparing Outcomes Using 1 Versus 2 Kirshner Wire Fixation in Patients With Severe Hallux Valgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 044/2568
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hallux Valgus Correction; Hallux Valgus; Hallux Valgus Deformity; Minimal Invasive Surgery
Keywords: DLMO; kirshner wire fixation; minimal invasive surgery
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixation with two kirshner wire in DLMO Surgery (Experimental): adding another kirshner wire through the osteotomized first metatarsal bone
  Interventions: Procedure: 2 Kirshner wire fixation
- fixation with one kirshner wire in DLMO surgery (No Intervention): using a standard technique of one kirshner wire fixation at first metatarsal bone

INTERVENTIONS:
Procedure: 2 Kirshner wire fixation — additional Kirshner wire fixation of first metatarsal bone
  Arms: fixation with two kirshner wire in DLMO Surgery

SUMMARY:
Comparing the radiographic and functional outcomes by using a Minimal invasive procedure to treat Hallux Valgus ; Distal linear Metatarsal Osteotomy -

1 Kirshner wire fixation versus two Kirshner wire fixation

DETAILED DESCRIPTION:
This is a randomise controlled trial between two groups patients, which are assigned to two different interventions, undergoing minimal invasive Hallux valgus surgery.

2nd generation of Minimal invasive surgery was selected in hallux valgus surgery due to its availability, cost effectiveness, reduced pain , and the overall simplicity of the operation, providing smaller surgical scars, and less op time , as well as blood loss.

this was done by making a osteotomy cut at the first metatarsal neck and placing one intramedullary Kirshner wire through the first metatarsal joint.

However the stability and the complication of this technique still remains - such as recurrence, K wire loosening, pin tract infection and malunion.

We believe that by adding another intramedullary Kirshner wire to fix the first metatarsal accoss the Metatarsophalangeal joint, the stability of the construct will improve and maintain a reduced hallux valgus angle ,and reduce the rate of complications , ultimately improving pain and functional outcome of the patient.

the participants were purposely randomized, and divided into two equal groups with 25 cases. the control group recieved a fixation with one Kirshner wire (standard) and the experimental group recieved a fixation with two Kirshner wire. Data were analyzed using paired T test , wilcoxon signed-rank test and chi squared test

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 year
* pain along medial surface of first MTP joint
* radiographic finding : medial deviation of first Metatarsal bone , and lateral deviation of Big toe
* complete a follow up period of 1 year , filling questionaires and undergone radiographic examination every visit
* radiographic finding : Hallux valgus angle >20 , Intermetatarsal angle > 10 degrees
* failed conservative treatment for atleast 8 months , with persistent pain along medial eminence and having difficulty walking, bearing weight

Exclusion Criteria:

* previous injury/fracture at big toe
* deviation/ subluxation of 1st MTP joint from traumatic event
* arthritic change of metatarsal bone, phalangeal bone of big toe
* previous/active infection , open wound along first metatarsal and big toe
* patient denied enrolling in study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Hallux Valgus Angle ( HVA ) | baseline, 2 week , 1 month , 2 month, 4 month , 8 month, 12 month
  degree of long axis of first Metatarsal to first proximal phalanx big toe

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Vadhana Memorial hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided